CLINICAL TRIAL: NCT03098797
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Crossover Trial to Evaluate the Safety and Efficacy of Subcutaneous Injections of Elamipretide in Subjects With Genetically Confirmed Barth Syndrome Followed by Open-Label Treatment
Brief Title: A Trial to Evaluate Safety, Tolerability and Efficacy of Elamipretide in Subjects With Barth Syndrome
Acronym: TAZPOWER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIBA-201
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Barth Syndrome
Keywords: Barth Syndrome; elamipretide; MTP-131; Stealth; Stealth BT; BTHS
MeSH Terms: conditions — Barth Syndrome | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Intervention Model Description: 28 weeks, double-blinded crossover followed by a 168-week open label long term safety & tolerability trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elamipretide, then Placebo (Experimental): Experimental Part 1: 12 weeks of single daily SC doses of 40 mg elamipretide in Treatment Period 1 followed by 12 weeks of treatment with placebo in Treatment Period 2 (separated by a 4 week washout period).
  Experimental Open Label Extension Part 2: All subjects will receive Elamipretide 40mg SC daily injections for up to 168 weeks
  Interventions: Drug: Elamipretide; Drug: Placebo
- Placebo , then Elamipretide (Placebo Comparator): Placebo Comparator Part 1: 12 weeks of single daily SC doses of placebo in Treatment Period 1 followed by 12 weeks of treatment with 40 mg elamipretide in Treatment Period 2 (separated by a 4 week washout period).
  Placebo Comparator Open Label Extension Part 2: All subjects will receive Elamipretide 40mg SC daily injections for up to 168 weeks
  Interventions: Drug: Elamipretide; Drug: Placebo

INTERVENTIONS:
Drug: Elamipretide — 40 mg daily subcutaneous injection for 12 weeks
  Other Names: MTP-131
Drug: Placebo — daily subcutaneous injection for 12 weeks
  Other Names: Placebo Comparator

SUMMARY:
A randomized, double-blind cross over trial to evaluate the safety, efficacy, and tolerability of elamipretide in subjects with Barth syndrome.

DETAILED DESCRIPTION:
A phase 2 randomized, double-blind, placebo-controlled crossover trial to evaluate the safety, tolerability, and efficacy of subcutaneous injections of elamipretide in subjects with genetically confirmed Barth syndrome followed by open-label treatment extension. Part 1 was a randomized, double-blind, placebo-controlled, crossover trial to assess safety, tolerability, and efficacy single daily subcutaneous (SC) doses of 40 mg elamipretide administered for 12 weeks in subjects with Barth syndrome. Part 2: This was an open-label extension trial to assess the long-term safety, tolerability, and longitudinal trends in efficacy single daily SC doses of 40 mg elamipretide for up to 192 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Barth Syndrome
* Male aged 12 and above
* At the screening visit, eGFR must meet the following:

  1. Body weight >30 kg AND eGFR ≥ 90mL/min at screening
  2. Body weight >40kg AND eGFR ≥60 but <90mL/min/ 1.73m² at screening
* Ambulatory and impaired during the baseline 6MWT
* On stable medication for 30 days prior to the baseline visit

Exclusion Criteria:

* Participated in another interventional clinical trial within 30 days of or is currently enrolled in a non-interventional clinical trial at the baseline visit potentially confounding with this trial
* Prior or current medical condition that would prevent the subject from safely participating in the trial
* Undergone any inpatient hospitalizations within 30 days of the baseline visit
* Is undergoing an apparent pubertal growth spurt
* Has uncontrolled hypertension
* History of substance abused within the year before the baseline visit or is likely to be uncompliant
* History of heart transplantation or current placement on the waiting list for a heart transplant
* For subjects with an ICD: known occurrence of ICD discharge in the 3 months prior to the baseline visit
* For subjects without an ICD: expected to undergo an implantation of an ICD during the conduct of the study
* Currently receiving treatment with chemotherapeutic agents or immunosuppressant agents or has received prior radiation therapy to the chest
* Recipient of stem cell or gene therapy or is currently being treated by a therapeutic investigational device

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Vernon, MD, PhD, Principal Investigator — McKusick-Nathans Institute of Genetic Medicine, Johns Hopkins University, Baltimore, MD, USA
Locations (1):
- McKusick-Nathans Institute of Genetic Medicine, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwaltney C, Shields A, Love E, Ollis S, Stokes J, Mazar I, Arenson E, Aiudi A, Wirth RJ, Houts C. Initial Psychometric Evaluation of the Barth Syndrome Symptom Assessment (BTHS-SA) for Adolescents and Adults in a Phase 2 Clinical Study. Orphanet J Rare Dis. 2025 Apr 25;20(1):199. doi: 10.1186/s13023-025-03693-5. PMID 40281531
- [Derived] Kim AY, Vernon H, Manuel R, Almuqbil M, Hornby B. Quality of life in Barth syndrome. Ther Adv Rare Dis. 2022 Jun 11;3:26330040221093743. doi: 10.1177/26330040221093743. eCollection 2022 Jan-Dec. PMID 37180415

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Elamipretide, Then Placebo: Part 1: Patients will be randomized to receive 12 weeks of elamipretide in one of the two treatment periods. All subjects will receive 12 weeks of elamipretide, 4 weeks of washout, then 12 weeks of placebo followed by a 4-week washout period before Part 2.
  Elamipretide: 40 mg daily subcutaneous injection for 12 weeks Placebo: subcutaneous injection for 12 weeks Part 2: Open Label Extension: Subjects are to be treated with daily 40 mg SC elamipretide for up to 192 weeks.
- Placebo, Then Elamipretide: Patients will be randomized to receive 12 weeks of placebo in one of the two treatment periods. All subjects will receive 12 weeks of placebo, followed by a 4 week washout period and then 12 weeks of elamipretide followed by a 4-week washout period before Part 2.
  Placebo: subcutaneous injection for 12 weeks Elamipretide: 40 mg daily subcutaneous injection for 12 weeks
  Part 2: Open Label Extension: Subjects are to be treated with 40 mg SC elamipretide for up to 192 weeks.
Period: First Intervention (12 Weeks)
Arm/Group | Experimental: Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Experimental: Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention (12 Weeks)
Arm/Group | Experimental: Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Part 2 Open Label Extension
Arm/Group | Experimental: Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 5 (Participants who received in Part 1 Elamipretide first, then Placebo. 1 participant declined to continue to Part 2) | 5 (Participants who in Part 1 received: Placebo first then Elamipretide. 1 participant declined to continue to Part 2)
Week 12 | 5 | 5
Week 36 | 3 | 5
Week 168 | 3 | 5
Completed | 3 | 5
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Elamipretide (Treatment AB): Patients will be randomized to receive 12 weeks of elamipretide in one of the two treatment periods. All subjects will receive 12 weeks of elamipretide, 4 weeks of washout, and 12 weeks of placebo and 4 weeks of follow up (for those not continuing to Part 2).
  Elamipretide: 40 mg daily subcutaneous injection for 12 weeks Placebo: daily subcutaneous injection for 12 weeks
- Experimental Placebo (Treatment BA): Patients will be randomized to receive 12 weeks of placebo in one of the two treatment periods. All subjects will receive 12 weeks of placebo, 4 weeks of washout, and 12 weeks of elamipretide, and 4 weeks of follow up (for those not continuing to Part 2).
  Placebo: daily subcutaneous injection for 12 weeks Elamipretide: 40 mg daily subcutaneous injection for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Experimental: Elamipretide (Treatment AB) | Experimental Placebo (Treatment BA) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All participants for whom Age was measured.
  years
    Part 1 | 23.3 (9.07) | 15.7 (3.33) | 19.5 (7.65)
    PART 2: OLE: number analyzed (Participants) | 5 | 5 | 10
    PART 2: OLE | 21.8 (9.23) | 16.2 (3.42) | 19.0 (7.20)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants for whom sex was measured.
  Participants
    Part 1: Female | 0 | 0 | 0
    Part 1: Male | 6 | 6 | 12
    Part 2 (OLE): number analyzed (Participants) | 5 | 5 | 10
    Part 2 (OLE): Female | 0 | 0 | 0
    Part 2 (OLE): Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All individuals for whom race was measured.
  Participants
    Part 1: American Indian or Alaska Native | 0 | 0 | 0
    Part 1: Asian | 0 | 0 | 0
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part 1: Black or African American | 0 | 0 | 0
    Part 1: White | 6 | 5 | 11
    Part 1: More than one race | 0 | 1 | 1
    Part 1: Unknown or Not Reported | 0 | 0 | 0
    Part 2 (OLE): number analyzed (Participants) | 5 | 5 | 10
    Part 2 (OLE): American Indian or Alaska Native | 0 | 0 | 0
    Part 2 (OLE): Asian | 0 | 0 | 0
    Part 2 (OLE): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part 2 (OLE): Black or African American | 0 | 0 | 0
    Part 2 (OLE): White | 5 | 4 | 9
    Part 2 (OLE): More than one race | 0 | 1 | 1
    Part 2 (OLE): Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: All participants for whom Body Mass Index was measured.
  kg/m^2
    Part 1 | 18.23 (3.677) | 16.88 (4.179) | 17.56 (3.818)
    Part 2 OLE: number analyzed (Participants) | 5 | 5 | 10
    Part 2 OLE | 18.14 (4.103) | 17.54 (4.313) | 17.84 (3.981)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Distance Walked During the 6-Minute Walk Test (6MWT) by Visit
Description: Average distance walked in meters during the 6-minute walk test (6MWT) at end of treatment, where end of treatment means end of Visit 5 (Week 12) for Period 1 and end of Visit 10 (Week 12) for Period 2. Results were pooled for each 12 week period.
Time Frame: Pre-dose to Week 12 (end of treatment)
Population: All participants for whom 6MWT was measured.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Experimental: Elamipretide: Subjects were randomized (in a ratio of 1:1) to one of two sequence groups:
  * Sequence 1: 12 weeks of single daily SC doses of 40 mg elamipretide in Treatment Period 1 followed by 12 weeks of treatment with placebo in Treatment Period 2 (separated by a 4-week washout period).
  * Sequence 2: 12 weeks of single daily SC doses of placebo in Treatment Period 1 followed by 12 weeks of treatment with 40 mg elamipretide in Treatment Period 2 (separated by a 4-week washout period).
- Placebo: Subjects were randomized (in a ratio of 1:1) to one of two sequence groups:
  * Sequence 1: 12 weeks of single daily SC doses of 40 mg elamipretide in Treatment Period 1 followed by 12 weeks of treatment with placebo in Treatment Period 2 (separated by a 4-week washout period).
  * Sequence 2: 12 weeks of single daily SC doses of placebo in Treatment Period 1 followed by 12 weeks of treatment with 40 mg elamipretide in Treatment Period 2 (separated by a 4-weekwashout period).
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
meters
  Pre-dose | 400.1 (55.07) | 412.6 (60.16)
  Week 12 (End of Treatment | 443.1 (65.43) | 443.9 (77.10)

2. Primary Outcome: Part 1: Total Fatigue Score Based on the BTHS-SA by Visit.
Description: Total Fatigue Score (Q1, Q2, and Q4) Based on the BarTH Syndrome Symptom Assessment (BTHS-SA) by visit at predose, Weeks 1, 4, 8, and 12 (end of treatment). The BTHS-SA is 3-question fatigue assessment using a 0 to 4-point scale for each question where no fatigue =0 and very severe fatigue =4, with scores from all 3 questions combined and averaged for all subjects; a lower score means better outcome, higher score means a worse outcome. Combined Min score=0, max score =12. Weekly values are based on the weekly average of the last 7 days before the site or visiting nurse visit for both periods. Results from each 12-week period were combined, where end of treatment for Period 1 =Visit 5 (week 12), and End of Period 2 = Visit 10 (week 12)
Time Frame: Pre-dose, Weeks 1, 4, 8, and 12 (end of treatment)
Population: All participants for whom Total Fatigue Score was measured
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Elamipretide; Placebo: Subjects were randomized (in a ratio of 1:1) to one of two sequence groups:
  * Sequence 1: 12 weeks of single daily SC doses of 40 mg elamipretide in Treatment Period 1 followed by 12 weeks of treatment with placebo in Treatment Period 2 (separated by a 4-week washout period).
  * Sequence 2: 12 weeks of single daily SC doses of placebo in Treatment Period 1 followed by 12 weeks of treatment with 40 mg elamipretide in Treatment Period 2 (separated by a 4-weekwashout period).
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale
  Pre-dose | 7.672 (1.9360) | 7.433 (1.3848)
  Week 1 | 6.837 (2.1114) | 6.994 (1.7093)
  Week 4: number analyzed (Participants) | 11 | 12
  Week 4 | 6.220 (2.3325) | 6.485 (1.4447)
  Week 8 | 6.089 (1.8344) | 6.196 (1.7815)
  Week 12: number analyzed (Participants) | 11 | 12
  Week 12 | 6.305 (2.0612) | 6.240 (1.6384)

3. Secondary Outcome: Part 2: Distance Walked During the 6MWT
Description: Change from baseline for distance walked in meters during the 6-minute walk test (6MWT) by visit where Baseline= Part 1 Period 1 Pre-dose
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96, 168, 192
Population: All participants for whom distance walked in 6MWT was measured.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Part 1: Elamipretide (Sequence AB): Part 2: Participants received treatment with 40 mg daily subcutaneous injection elamipretide for up to 192 weeks.
- Part 2: Placebo (Sequence BA): Part 2: Participants were treated with daily 40 mg daily subcutaneous injection elamipretide for up to 192 weeks.
Arm/Group | Part 1: Elamipretide (Sequence AB) | Part 2: Placebo (Sequence BA)
Number analyzed (Participants) | 5 | 5
meters
  Part 2: Week 12 | 45.4 (55.73) | 75.6 (87.25)
  Part 2: Week 24: number analyzed (Participants) | 4 | 5
  Part 2: Week 24 | 79.8 (23.54) | 100.4 (94.61)
  Part 2: Week 36: number analyzed (Participants) | 3 | 5
  Part 2: Week 36 | 68.0 (31.19) | 112.6 (119.35)
  Part 2: Week 48: number analyzed (Participants) | 3 | 5
  Part 2: Week 48 | 87.3 (25.58) | 103.4 (102.02)
  Part 2: Week 72: number analyzed (Participants) | 3 | 5
  Part 2: Week 72 | 121.7 (20.74) | 97.8 (117.53)
  Part 2: Week 96: number analyzed (Participants) | 1 | 3
  Part 2: Week 96 | 128.0 | 63.7 (69.14)
  Part 2: Week 168: number analyzed (Participants) | 3 | 5
  Part 2: Week 168 | 89.3 (32.75) | 100.2 (78.10)
  Part 2: Week 192: number analyzed (Participants) | 1 | 2
  Part 2: Week 192 | 118.0 | 125.0 (28.28)

4. Secondary Outcome: Part 2: Change From Baseline: Total Fatigue Score (Q1, Q2, and Q4) Based on the BTHS-SA by Visit
Description: Change from Baseline (mean) in Total Fatigue Score (Q1, Q2, and Q4) Based on the BarTH Syndrome Symptom Assessment (BTHS-SA) by visit. The BTHS-SA is 3-question fatigue assessment using a 0-4 point scale for each question where no fatigue =0 and very severe fatigue =4, with scores from all 3 questions combined and averaged for all subjects by visit; a lower score means better outcome, higher score means a worse outcome. Change from baseline: an increase in scores would mean worse outcome, a decrease in scores means better outcome. Combined Min score=-12, max score =12. Weekly values are based on the weekly average of the last 7 days before the site or visiting nurse visit for both periods. Baseline= Period 1 Predose.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96, 120, 144, 168, 192
Population: All participants for whom Total Fatigue Score was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 2: OLE: (Treatment AB): Part 2: Participants received treatment with 40 mg SC elamipretide for up to 192 weeks.
- Part 2: OLE: (Treatment BA): Part 2: Participants were treated with daily 40 mg SC elamipretide for up to 192 weeks.
Arm/Group | Part 2: OLE: (Treatment AB) | Part 2: OLE: (Treatment BA)
Number analyzed (Participants) | 5 | 5
score on a scale
  Baseline | -2.425 (2.0849) | -1.540 (1.3653)
  Week 12 | -1.800 (2.4838) | -1.314 (1.4237)
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | -1.500 (2.0253) | -0.314 (1.0816)
  Week 36: number analyzed (Participants) | 3 | 5
  Week 36 | -2.667 (3.6821) | -1.714 (1.0583)
  Week 48: number analyzed (Participants) | 3 | 5
  Week 48 | -1.000 (2.9172) | -0.314 (1.0650)
  Week 72: number analyzed (Participants) | 3 | 5
  Week 72 | -2.667 (3.4827) | -1.114 (1.1301)
  Week 96: number analyzed (Participants) | 2 | 3
  Week 96 | -3.500 (2.5254) | -0.357 (1.5763)
  Week 120: number analyzed (Participants) | 3 | 5
  Week 120 | -3.000 (2.9172) | -0.114 (1.0309)
  Week 144: number analyzed (Participants) | 3 | 5
  Week 144 | -2.667 (2.2961) | -0.314 (2.0067)
  Week 168: number analyzed (Participants) | 3 | 5
  Week 168 | -2.333 (4.0515) | -0.514 (0.7309)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | -5.286 | -1.107 (0.5556)

5. Secondary Outcome: Part 1: Muscle Strength as Measured by HHD by Visit
Description: Muscle strength as measured by handheld dynamometry (HHD) in Newtons, where end of treatment means end of Visit 5 (Week 12) for Period 1 and end of Visit 10 (Week 12) for Period 2. Results were pooled for each 12 week period. Handheld dynamometry assesses the average strength of the knee extensors of both legs.
Time Frame: Pre-dose to Week 12 (end of treatment)
Population: All participants for whom muscle strength as measured by handheld dynamometry was measured.
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
Newtons
  Pre-dose | 131.236 (29.9004) | 123.100 (24.6762)
  Week 12 | 135.934 (52.2796) | 129.253 (34.2395)

6. Secondary Outcome: Part 2: Change From Baseline: Muscle Strength by HHD (Newtons) by Visit
Description: Muscle strength as measured by handheld dynamometry (HHD) in Newtons. Handheld dynamometry assesses the average strength of the knee extensors of both legs. Change from baseline where Baseline= Part 1 Period 1 Pre-dose: the greater positive change, the better the outcome, the smaller positive change (or negative change) the number the worse the outcome.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96,168, 192
Population: All participants for whom Muscle Strength by HHD (Newtons) was measured.
Measure: Mean (Standard Deviation); unit: Newtons
Groups:
- Part 2: OLE: (Treatment AB): Part 2: Participants received treatment with 40 mg daily subcutaneous injection elamipretide for up to 192 weeks.
- Part 2: OLE: (Treatment BA): Part 2: Participants were treated with daily 40 mg daily subcutaneous injection elamipretide for up to 192 weeks.
Arm/Group | Part 2: OLE: (Treatment AB) | Part 2: OLE: (Treatment BA)
Number analyzed (Participants) | 5 | 5
Newtons
  Week 12 | 33.606 (24.7304) | 42.147 (34.9498)
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | 54.073 (29.7699) | 54.068 (37.3060)
  Week 36: number analyzed (Participants) | 3 | 5
  Week 36 | 68.798 (22.8892) | 48.351 (31.1331)
  Week 48: number analyzed (Participants) | 3 | 5
  Week 48 | 69.613 (20.8788) | 45.704 (56.8895)
  Week 72: number analyzed (Participants) | 3 | 5
  Week 72 | 62.089 (33.4753) | 32.071 (31.7087)
  Week 96: number analyzed (Participants) | 1 | 3
  Week 96 | 93.745 | 38.848 (18.1422)
  Week 168: number analyzed (Participants) | 3 | 5
  Week 168 | 57.751 (17.7509) | 61.897 (19.1573)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | 42.368 | 32.140 (17.9287)

7. Secondary Outcome: Part 1: 5XSST by Visit
Description: Time (in seconds) to complete the Five Times Sit-To-Stand, where end of treatment means end of Visit 5 (Week 12) for Period 1 and end of Visit 10 (Week 12) for Period 2. Results were pooled for each 12 week period.
Time Frame: Pre-dose to Week 12 (end of treatment)
Population: All participants for whom 5XSST was measured.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
seconds
  Pre-dose: number analyzed (Participants) | 11 | 12
  Pre-dose | 12.965 (3.3366) | 13.710 (5.3088)
  Week 12 | 14.023 (5.4508) | 13.749 (6.1024)

8. Secondary Outcome: Part 2: Change From Baseline: 5X Sit to Stand by Visit
Description: Change in baseline in time (in seconds), where Baseline= Part 1 Period 1 Pre-dose to complete the Five Times Sit-To-Stand by visit. More time means worse outcome, less time means better outcome.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96, 168, 192
Population: All participants for whom 5X Sit to Stand was measured.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Part 2: OLE: (Sequence AB): Part 2: Participants received treatment with 40 mg daily subcutaneous injection elamipretide for up to 192 weeks.
- Part 2: OLE: (Sequence BA): Part 2: Participants were treated with daily 40 mg daily subcutaneous injection elamipretide for up to 192 weeks.
Arm/Group | Part 2: OLE: (Sequence AB) | Part 2: OLE: (Sequence BA)
Number analyzed (Participants) | 5 | 5
seconds
  End of Part 1: number analyzed (Participants) | 4 | 5
  End of Part 1 | -0.773 (2.5323) | 0.400 (2.7824)
  Week 12: number analyzed (Participants) | 4 | 5
  Week 12 | -1.505 (2.1843) | 0.384 (3.7167)
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | -2.533 (2.7507) | -1.160 (2.8668)
  Week 36: number analyzed (Participants) | 3 | 5
  Week 36 | -3.700 (3.7649) | -0.344 (2.7035)
  Week 48: number analyzed (Participants) | 3 | 5
  Week 48 | -4.780 (2.9820) | -0.082 (2.6625)
  Week 72: number analyzed (Participants) | 3 | 5
  Week 72 | -4.770 (3.2043) | -0.454 (1.6369)
  Week 96: number analyzed (Participants) | 1 | 3
  Week 96 | -8.060 | -0.397 (3.6036)
  Week 168: number analyzed (Participants) | 3 | 5
  Week 168 | -4.320 (4.0307) | -0.986 (2.1857)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | -6.850 | -0.390 (1.5839)

9. Secondary Outcome: Part 1: SWAY Application Balance Assessments by Visit
Description: SWAY application balance assessment consists of five stances each performed for 10 seconds and scores postural stability on a scale from 0-100 with higher scores indicating better postural stability from Pre-dose to Week 12 (end of treatment), where end of treatment means end of Visit 5 (Week 12) for Period 1 and end of Visit 10 (Week 12) for Period 2. Results were pooled for each 12 week period.
Time Frame: Pre-dose to Week 12 (end of treatment)
Population: All participants for who SWAY application balance was measured.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
Score on a scale
  Pre-dose | 70.752 (19.7199) | 68.820 (24.7478)
  Week 12 | 78.698 (15.1554) | 71.353 (20.2515)

10. Secondary Outcome: Part 2: Change From Baseline: SWAY Application Balance Assessment
Description: Change from Baseline: SWAY Application Balance Assessment,where Baseline= Part 1 Period 1 Pre-doseSWAY application balance assessment consists of five stances each performed for 10 seconds and scores postural stability on a scale from 0-100 with higher scores indicating better postural stability. An increase from baseline is a better outcome and a decrease in score is a worse outcome.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96,168, 192
Population: All participants for whom SWAY Application Balance Assessment was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: OLE: (Sequence AB) | Part 2: OLE: (Sequence BA)
Number analyzed (Participants) | 5 | 5
score on a scale
  Week 12 | -3.152 (29.8419) | 10.464 (19.1971)
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | 12.190 (9.6799) | 6.664 (9.5896)
  Week 36: number analyzed (Participants) | 3 | 5
  Week 36 | 0.807 (14.9493) | 9.484 (11.3834)
  Week 48: number analyzed (Participants) | 3 | 5
  Week 48 | 5.773 (7.8814) | 15.260 (16.2540)
  Week 72: number analyzed (Participants) | 3 | 5
  Week 72 | 10.420 (1.7501) | 15.240 (14.3557)
  Week 96: number analyzed (Participants) | 1 | 3
  Week 96 | 12.840 | 18.433 (21.3323)
  Week 168: number analyzed (Participants) | 3 | 5
  Week 168 | 21.127 (14.1854) | 19.644 (18.6821)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | 15.100 | 13.080 (16.3483)

11. Secondary Outcome: Part 1: Patient Global Impression Scales of Symptoms
Description: Patient-reported health status over the past week, by visit, where end of treatment means end of Visit 5 (Week 12) for Period 1 and end of Visit 10 (Week 12) for Period 2. Results were pooled for each 12 week period. Scores range from 0-40 for adolescents and 0-50 for adults. PGI Scale is as follows: 0=None, 1=Mild, 2=Moderate, 3=Severe, and 4=Very Severe. Higher score means worse health status, means worse outcome; lower score means better health status, means better outcome.
Time Frame: Pre-dose, Week 1, Week 12 (end of treatment)
Population: All participants for whom Patient Global Impression Scales of Symptoms was measured.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
Score on a scale
  Predose | 1.7 (0.65) | 1.8 (0.83)
  Week 1 | 1.7 (0.89) | 1.5 (1.00)
  Week 12 | 1.4 (0.79) | 1.6 (0.67)

12. Secondary Outcome: Part 2: Change From Baseline: Patient Global Impression Scales of Symptoms by Visit
Description: Part 2: Change from Baseline: Patient Global Impression Scales of Symptoms by Visit Patient-reported health status over the past week where Baseline= Part 1 Period 1 Pre-dose, administered at Week 12 for Period 1 and Period 2. Scores range from 0-40 for adolescents and 0-50 for adults. PGI Scale is as follows: 1=None, 2=Mild, 3=Moderate, 4=Severe, and 5=Very Severe. Change from baseline: Higher score means worse health status, means worse outcome; lower score means better health status, means better outcome.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96, 120, 144, 168, 192
Population: All participants for whom Patient Global Impression Scales of Symptoms was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: OLE: (Sequence AB) | Part 2: OLE: (Sequence BA)
Number analyzed (Participants) | 5 | 5
score on a scale
  End of Part 1 | 0.0 (0.00) | -0.4 (0.55)
  Week 12 | -0.2 (1.10) | -0.6 (0.55)
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | -0.3 (0.50) | -0.4 (0.55)
  Week 36: number analyzed (Participants) | 3 | 5
  Week 36 | -0.7 (1.15) | -0.6 (0.55)
  Week 48: number analyzed (Participants) | 3 | 5
  Week 48 | -0.7 (1.15) | 0.0 (0.00)
  Week 72: number analyzed (Participants) | 3 | 5
  Week 72 | -0.7 (1.15) | -0.4 (0.55)
  Week 96: number analyzed (Participants) | 2 | 3
  Week 96 | -0.5 (2.12) | -0.3 (0.58)
  Week 120: number analyzed (Participants) | 3 | 5
  Week 120 | -0.7 (1.15) | -0.6 (0.55)
  Week 144: number analyzed (Participants) | 2 | 5
  Week 144 | -1.0 (1.41) | -0.8 (0.45)
  Week 168: number analyzed (Participants) | 3 | 5
  Week 168 | -0.7 (1.15) | -0.6 (0.55)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | -2.0 | -0.5 (0.71)

13. Secondary Outcome: Part 1: Part 1: Clinician Global Impression
Description: Clinician Global Impression Scale by visit: Clinician-reported overall health status at end of treatment, administered at Week 12 for Period 1 and Period 2. Scores range from 0-6 for both adolescents and adults. PGI Scale is as follows: 1= Very much Better, 2= Moderately Better, 3= A Little Better, 4= No Change, and 5= A Little Worse 6= Very much Worse. Higher score means worse health status, means worse outcome; lower score means better health status, means better outcome. End of treatment means end of Visit 5 (Week 12) for Period 1 and end of Visit 10 (Week 12) for Period 2. Results were pooled for each 12 week period.
Time Frame: Pre-dose to Week 12 (end of treatment)
Population: All participants for whom Patient Global Impression Scales of Symptoms was measured.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Experimental: Elamipretide | Placebo
Number analyzed (Participants) | 12 | 12
Score on a scale
  Predose | 1.8 (0.45) | 1.4 (0.51)
  12 weeks | 1.6 (0.51) | 1.6 (0.51)

14. Secondary Outcome: Part 2: Change From Baseline: CGI Symptom Scale
Description: Change from Baseline: CGI Symptom Scale by visit where Baseline= Part 1 Period 1 Pre-dose. Clinician Global Impression Scale: Clinician-reported overall health status at end of treatment, administered at Week 12 for Period 1 and Period 2. Scores range from 0-6 for both adolescents and adults. PGI Scale is as follows: 1= Very much Better, 2= Moderately Better, 3= A Little Better, 4= No Change, and 5= A Little Worse 6= Very much Worse. Change from baseline: higher score means worse health status, means worse outcome; lower score means better health status, means better outcome.
Time Frame: Baseline to Weeks 12, 24, 36, 48, 72, 96, 120, 144, 168, 192
Population: All participants for whom Patient Global Impression Scales of Symptoms was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: OLE: (Sequence AB) | Part 2: OLE: (Sequence BA)
Number analyzed (Participants) | 5 | 5
score on a scale
  Week 12 | -0.4 (0.55) | 0.0 (0.00)
  Week 24: number analyzed (Participants) | 4 | 5
  Week 24 | -1.3 (0.96) | -0.4 (0.55)
  Week 36: number analyzed (Participants) | 3 | 5
  Week 36 | -1.3 (0.58) | -0.2 (0.84)
  Week 48: number analyzed (Participants) | 3 | 5
  Week 48 | -1.3 (0.58) | -0.4 (0.55)
  Week 72: number analyzed (Participants) | 3 | 5
  Week 72 | -1.3 (0.58) | -0.6 (0.55)
  Week 96: number analyzed (Participants) | 2 | 3
  Week 96 | -1.0 (0.00) | -0.7 (0.58)
  Week 120: number analyzed (Participants) | 3 | 5
  Week 120 | -1.7 (0.58) | -1.0 (0.71)
  Week 144: number analyzed (Participants) | 3 | 5
  Week 144 | -1.3 (0.58) | -0.6 (0.55)
  Week 168: number analyzed (Participants) | 3 | 5
  Week 168 | -1.3 (0.58) | -0.8 (0.84)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | -1.0 | -1.5 (0.71)

ADVERSE EVENTS:
Time Frame: Part 1: Participants were followed for a total of 28 weeks, they had a treatment period for 12 weeks, a washout period of 4 weeks, then another treatment period of 4 weeks. Part 2 OLE: Participants who agreed to proceed to Part 2 were followed for up to 192 weeks.
Groups:
- Part 2 (OLE): Elamipretide (Sequence AB): Part 2: Participants from Part 1 who received 12 weeks of elamipretide first, placebo for the last 12 weeks of treatment, then proceeded to Part 2 OLE and received up to 192 weeks of daily subcutaneous injections of 40mg elamipretide.
- Part 2 (OLE): Elamipretide (Sequence BA): Part 2: Participants from Part 1 who received 12 weeks of placebo first, then elamipretide for the last 12 weeks of treatment, then proceeded to Part 2 OLE and received up to 192 weeks of daily subcutaneous injections of 40mg elamipretide.
- Part 1: Elamipretide: Participants who received Elamipretide either in the first or last 12 weeks of treatment.
- Part 1: Placebo: Participants who received Placebo either in the first or last 12 weeks of treatment.
Arm/Group | Part 2 (OLE): Elamipretide (Sequence AB) | Part 2 (OLE): Elamipretide (Sequence BA) | Part 1: Elamipretide | Part 1: Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/5 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 2 (OLE): Elamipretide (Sequence AB) (N=5) | Part 2 (OLE): Elamipretide (Sequence BA) (N=5) | Part 1: Elamipretide (N=12) | Part 1: Placebo (N=12)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Mucositis (General disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Abscess of Right Axilla (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 2 (OLE): Elamipretide (Sequence AB) (N=5) | Part 2 (OLE): Elamipretide (Sequence BA) (N=5) | Part 1: Elamipretide (N=12) | Part 1: Placebo (N=12)
Injection site bruising (General disorders) | 0 | 1 | 3 | 0
Medical site device erythema (General disorders) | 0 | 0 | 1 | 1
Medical device site irritation (General disorders) | 0 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Injection site erythema (General disorders) | 3 | 5 | 12 | 3
Injection site pruritus (General disorders) | 3 | 5 | 8 | 2
Injection site pain (General disorders) | 3 | 4 | 9 | 4
Injection site induration (General disorders) | 2 | 3 | 8 | 2
Injection site urticaria (General disorders) | 2 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 5 | 1 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 1 | 3
Weight decreased (Investigations) | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Administration site pain (General disorders) | 0 | 0 | 0 | 1
Injection site erosion (General disorders) | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 1
Injection site scab (General disorders) | 0 | 1 | 1 | 0
Medical device site pruritus (General disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 1
Pneumonia chlamydial (Infections and infestations) | 0 | 0 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Left ventricular dilatation (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0
Injection site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0
Echocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 1 | 0 | 0
Lymph node palpable (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 0 | 0
Vaccination site rash (General disorders) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT03098797/Prot_SAP_000.pdf